CLINICAL TRIAL: NCT05428254
Title: The Effectiveness of Capacitive and Resistive Radiofrequency Therapy Alone or With Manual Therapy in the Treatment of Patients With Chronic Non-specific Mechanical Neck Pain.
Brief Title: Radiofrequency Therapy for Chronic Neck Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Umm Al-Qura University (Other)
Collaborators: Deanship of scientific research at Umm Al-Qura university (Unknown)
Responsible Party: Principal Investigator, Mohamed Alayat, Associate Professor of Physical Therapy, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-MED-06-1111
Record Dates: First submitted 2022-06-12; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Neck Pain, Posterior
MeSH Terms: conditions — Neck Pain | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: A total of 60 patients will participle in the study. They will be recruited from the hospital in Mecca, Saudi Arabia. They will be randomized into three groups. Group I will be treated with stretching exercises (EX) and manual therapy (Manual + EX group). Group II will be treated with CRRT plus EX without manual therapy (CRRT+ EX group). Group III will be treated by EX plus manual therapy applied during CRRT for groups (Manual + CRRT+ EX group). For group II and III, capacitive electrodes will be applied for five minutes. Then the resistive electrodes will be applied for 10 minutes and finally the capacitive will be applied again for another five minutes.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Individuals with non-specific CNP will be evaluated and referred by independent physicians from orthopedic department at Makkah hospitals. The first author will conduct the processes of participant enrollment and allocation. The allocation of patients is blinded to the assessor and to the therapist. By sealed envelopes, the allocation concealment is achieved. All participants will be eligible to participate after evaluation of independent physician. The physician conducts the processes of participant enrollment, and allocation. The same therapist will treat the patients and the study variables is measured by the same assessors. Randomization is performed using online GraphPad and creating a random number for each patient. Neither the assessor nor the CRRT applicant is oriented about the randomization process. The same therapist will treat the patients, and the study variables will be measured by the same assessor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise and Manual therapy (Active Comparator): Group I will be treated with stretching exercises (EX), manual therapy (EX group) and serves as a control group.
  Stretching of the neck extensor, upper fibers of trapezius, levator scapulae and scalenus muscles. stretching is applied for at least 15 seconds and repeated ten times in each session. Mobilization of the facet joint of the cervical vertebrae is performed after neck exercises.
  Interventions: Other: Exercise therapy
- Exercise and radiofrequency therapy (Active Comparator): Group II will be treated with capacitive and resistive radiofrequency therapy plus EX without manual therapy (CRRT+ EX group).
  In addition to neck stretching exercises, they will receive 20 minutes of CRRT. Both the capacitive and resistive electrodes. CRRT is applied by the INDIBA radiofrequency therapy. INDIBA radiofrequency therapy has a long wavelength diathermy with frequency of 488 KHz range. The integration of two operational modes capacitive electrode (CAP) and (RES), makes it possible to combine sub-thermal (electric) and thermal effects. Indiba radiofrequency has output frequency: 448kHz ± 1 kHz with Maximum output power in RES mode: 100 W and in CAP mode: 350 VA. Capacitive electrodes will be applied for five minutes. Then the resistive electrodes will be applied for 10 minutes and finally the capacitive will be applied again for another five minutes.
  Interventions: Other: Capacitive and Resistive Radiofrequency therapy; Other: Exercise therapy
- Exercise, Manual and Radiofrequency therapy (Active Comparator): Patients in this group will receive the same program of exercises as in group one. in addition, patients will receive the CRRT as in group two and the mobilization of the facet joints of the cervical vertebrae is applied while applied the CRRT by a trained physiotherapist. The same protocol of mobilization is applied for group one and three.
  Interventions: Other: Capacitive and Resistive Radiofrequency therapy; Other: Exercise therapy

INTERVENTIONS:
Other: Capacitive and Resistive Radiofrequency therapy — TECAR or CRRT is electromagnetic waves produced by high frequency electrical current that are able to penetrate very deep and produce a long-lasting heat which stimulates the superficial and dep tissues and produce a potent long-lasting pain-relieving effect. Mild intensity of heat produced by the long wave diathermy may be used to promote proliferation (Hernández-Bule et al., 2014) and improve the vascularization of skin and muscles.
  The integration of two operational modes, Capacitive (CAP) and Resistive (RES), makes it possible to combine sub-thermal (electric) and thermal effects. Indiba radiofrequency has output frequency: 448kHz ± 1 kHz with Maximum output power in RES mode: 100 W and in CAP mode: 350 VA. The capacitive used an isolated metal coated electrode acts as a dielectric surface which concentrate the electrical charges near the capacitive electrode While the resistive electrode causing the diffusion of electrical charges which accumulate near bone and soft tissues.
  Other Names: Transfer Electrical Capacitive And Resistive (TECAR therapy)
  Arms: Exercise and radiofrequency therapy; Exercise, Manual and Radiofrequency therapy
Other: Exercise therapy — Stretching of the neck extensor, upper fibers of trapezius, levator scapulae and scalenus muscles. stretching is applied for at least 15 seconds and repeated ten times in each session.

SUMMARY:
Background: Chronic neck pain (CNP) is a major health problem affecting individuals with high prevalence and subsequent complications which interfere with the physical, personnel, and psychological status. The capacitive and resistive radiofrequency therapy (CRRT) is a relatively new treatment modality used in rehabilitation with no evidence on its efficacy on chronic neck pain.

Objective: The aim of the present study is to investigate the effect of the CRRT alone or with manual therapy in the treatment of patients with patients with non-specific CNP.

Hypotheses Is the application of the CRRT when applied alone or with combination with manual therapy and exercises effective in decreasing pain and improving the function and strength in patients with non-specific chronic neck pain?? Methods: 60 patients will participle in the study. They will be recruited from the hospital in mecca, Saudi Arabia. They will be randomized into three groups. Group I will be treated with stretching exercises (EX) and manual therapy (Manual + EX group). Group II will be treated with CRRT plus exercises (CRRT+ EX group). Group III will be treated by EX plus manual therapy applied during CRRT for groups (Manual + CRRT+ EX group). For groups II and III, capacitive electrodes will be applied for five minutes. Then the resistive electrodes will be applied for 10 minutes and finally the capacitive will be applied again for another five minutes. Assessment of the neck pain, function, CROM, trigger points, neck muscle strength as well as neck angles will be performed. Measurement will be performed before, after 6 weeks, and 6 months of treatment as follow up measurements. Multivariate analysis of variance was used to compare between and within groups. The level of statistical significance is set as P<0.05.

DETAILED DESCRIPTION:
Chronic neck pain (CNP) is a major health problem affecting individuals with high prevalence 90.4 to 86.8% of the population) and comes secondary to low back pain. It exerts negative pressure on personnel, their families, and health organizations in addition to the decreases of workdays and productivity loss. CNP may be associated with referred pain, restricted range of motion, headache, presence of trigger points, dysfunction of the cervical musculature and presence of faulty posture.

Rehabilitation of patients with CNP may include the mechanical, electrical and /or, thermal modalities which are applied with the manual techniques and exercise therapy. The capacitive and resistive radiofrequency therapy (CRRT) is a long-wave diathermy with a long-lasting thermal effect used to decrease pain and muscle spasm in case of lumbago, fibromyalgia, and knee osteoarthritis.

Literature comparing the efficacy of each modality with exercise or with manual therapy. Previous literature used CRRT for only its thermal effect. The CRRT may combine the effect of thermal, electrical, and mechanical modalities as well as the effect of exercise and manual therapy with a new technique not used previously. This study is the first study using CRRT with a new technique which combines the effect of the CRRT with the manual therapy to treat patients with CNP.

Objective of the project:

The aim of the present study is to investigate the effect of the CRRT in the treatment of patients with non-specific CNP. The CRRT will be applied to the posterior neck and shoulder areas for two sessions per week for six weeks. CRRT will be applied alone or combined with manual therapy and stretching exercises.

1. To investigate the short-term effect of the CRRT on the neck pain, function, and cervical range of motion (ROM), the pressure pain threshold of the trigger points trapezius upper fibers, neck muscle strength, and the neck angles.
2. Compare the effect of CRRT alone to the combined effect of CRRT and manual therapy on the measured outcomes.
3. To investigate the long-term effect of CRRT alone or combined with manual therapy on patients with non-specific CNP.

Hypotheses Is the application of the CRRT when applied alone or in combination with manual therapy and exercises effective in decreasing pain and improving the function and strength in patients with non-specific chronic neck pain??

Ethical Approval:

this protocol had an ethical approval from the Institute Review Board of biomedical research ethics committee, Umm Al-Qura University Makkah, Saudi Arabia A written consent form also will be provided for all participants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic neck pain.
2. Age is above 18 years.
3. patients had chronic pain ≥ 3 months,
4. The radiological examination showed that the patients is free from any discogenic cause of pain.
5. Patients are willing to stop medications.
6. Patients accepted to assign informed consent to participate in the current study and will attend the lab twice a week for six successive weeks.

Exclusion Criteria:

1. They have any known significant medical conditions such as hypertension, asthma, cardiac disease, or systemic disease that adversely affect them during testing.
2. Previous neck surgery/injection for the last six months.
3. Previous vertebral fracture or malignancy.
4. Patients have a discogenic pain or any other radicular manifestation to the upper limb.
5. Unable to commit study requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Measurement will be performed before treatment.
  The pain will be measured using a visual analogue scale (VAS). This scale is a 10-centimeter drawn line.
Pain intensity | Measurement will be performed after 6 weeks of treatment.
  The pain will be measured using a visual analogue scale (VAS). This scale is a 10-centimeter drawn line.
Pain intensity | Measurement will be performed after 3 months of treatment as follow up measurement.
  The pain will be measured using a visual analogue scale (VAS). This scale is a 10-centimeter drawn line.
Pain intensity | Measurement will be performed after 6 months of treatment as follow up measurement.
  The pain will be measured using a visual analogue scale (VAS). This scale is a 10-centimeter drawn line.

SECONDARY OUTCOMES:
Neck disability index | Measurement will be performed before treatment.
  The level of function is measured by the neck disability index. An Arabic version of neck disability index (NDI) will be filled for all patients. NDI is the most frequently functional activity index used for neck related disabilities and is considered as a valid and reliable measure used in patients with neck pain. NDI is a self-perceived disability neck pain from. Every patient is asked to mark the in each section which most describes his level of disability. Each item is recorded out of 5 for a maximum total score of 50
Neck disability index | Measurement will be performed after 6 weeks of treatment.
  The level of function is measured by the neck disability index. An Arabic version of neck disability index (NDI) will be filled for all patients. NDI is the most frequently functional activity index used for neck related disabilities and is considered as a valid and reliable measure used in patients with neck pain. NDI is a self-perceived disability neck pain from. Every patient is asked to mark the in each section which most describes his level of disability. Each item is recorded out of 5 for a maximum total score of 50
Neck disability index | Measurement will be performed after 3 months of treatment as a follow up measurement.
  The level of function is measured by the neck disability index. An Arabic version of neck disability index (NDI) will be filled for all patients. NDI is the most frequently functional activity index used for neck related disabilities and is considered as a valid and reliable measure used in patients with neck pain. NDI is a self-perceived disability neck pain from. Every patient is asked to mark the in each section which most describes his level of disability. Each item is recorded out of 5 for a maximum total score of 50
Neck disability index | Measurement will be performed after 6 months of treatment as a follow up measurement.
  The level of function is measured by the neck disability index. An Arabic version of neck disability index (NDI) will be filled for all patients. NDI is the most frequently functional activity index used for neck related disabilities and is considered as a valid and reliable measure used in patients with neck pain. NDI is a self-perceived disability neck pain from. Every patient is asked to mark the in each section which most describes his level of disability. Each item is recorded out of 5 for a maximum total score of 50

OTHER OUTCOMES:
Pressure pain threshold | Measurement will be performed before treatment.
  Trigger points in the posterior neck and upper fibers of trapezius muscle will be allocated and evaluated using the pressure algometer.
Pressure pain threshold | Measurement will be performed after 6 weeks of treatment.
  Trigger points in the posterior neck and upper fibers of trapezius muscle will be allocated and evaluated using the pressure algometer.
Pressure pain threshold | Measurement will be performed after 3 months of treatment as a follow up measurement.
  Trigger points in the posterior neck and upper fibers of trapezius muscle will be allocated and evaluated using the pressure algometer.
Pressure pain threshold | Measurement will be performed after 6 months of treatment as follow up measurement.
  Trigger points in the posterior neck and upper fibers of trapezius muscle will be allocated and evaluated using the pressure algometer.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Alayat, Ph.D., Principal Investigator — Umm Al-Qura University
Locations (1):
- Umm Al-Qura University, Faculty of Applied Medical Science, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided